CLINICAL TRIAL: NCT03611231
Title: Chidamide Maintenance Treatment After Autologous Hematopoietic Stem Cell Transplantation in Patients With Relapsed, Refractory or High-risk Lymphoma : a Prospective, Multi-centric, Single Arm, Open Label Phase II Clinical Trial
Brief Title: Chidamide Maintenance After Autologous Hematopoietic Stem Cell Transplantation for Relapsed, Refractory or High-risk Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Peking University International Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q06
Record Dates: First submitted 2018-06-25; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Experimental Tumor
MeSH Terms: conditions — Neoplasms, Experimental | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): chidamide
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide 20mg orally BIW. Treatment cycles are repeated every 4 weeks.
  Other Names: epidaza

SUMMARY:
Chidamide Maintenance Treatment After Autologous Hematopoietic Stem Cell Transplantation in Patients With Relapsed, Refractory or High-risk Lymphoma : a Prospective, Multi-centric, Single Arm, Open Label Phase II Clinical Trial

DETAILED DESCRIPTION:
Chidamide，a novel histone deacetylase inhibitor has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China. The aim of this study was to observe the efficacy and safety of Chidamide as Maintenance Treatment After Autologous Hematopoietic Stem Cell Transplantation in Patients With Relapsed, Refractory or High-risk Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients with B-NHL,NK/T-NHL and HL were confirmed by histopathology examination had received autologous hematopoietic stem cell transplantation (including secondary transplantation). Transplantation interval was 6-8 weeks before in the study. The first diagnostic risk classification or pre-transplant disease status of each type of lymphoma is as follows: 1)B-NHL: patients who are at high risk according to the corresponding international prognostic index in the first diagnosis(IPI>3 /aa IPI >2 /FLIPI>3); Patients must have received at least one first-line induction therapy but did not achieve CR or had relapse after CR; 2)NK/T-NHL: Including all patients, unlimited risk classification and pre-transplant disease status; 3)HL: Patients must have received at least one first-line induction therapy
2. Age 18-70 years, male or female;
3. ECOG performance status 0-1;
4. Organ function should fit the following : Renal function with serum creatinine < 160μmol/L; Liver function with Total bilirubin ≤2 times of normal maximum, ALT and AST≤3 times of normal maximum. Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusing capacity of lung for carbon monoxide (DLCO) ≥ 50% of expected corrected for hemoglobin. Adequate cardiac function with left ventricular ejection fraction ≥ 50%. No symptomatic cardiac disease;
5. Blood routine test: absolute neutrophil count ≥1.5×109/L, platelet ≥75×109/L, Hb ≥ 90g/L;
6. Life expectancy no less than 3 months;
7. Patients willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Patients relapsed after ASCT
2. Patients with HBsAg positive or HBcAb positive patients also detected HBV-DNA copy number positive;
3. Patients with active HCV infection;
4. Patients with active HIV infection;
5. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulopathy, connective tissue disease, severe infectious diseases and others;
6. Patients with liver cirrhosis or evidence of liver fibrosis;
7. Patients with a QTc longer than 500 ms;
8. Patients with mental disorders or those do not have the ability to consent;
9. Patients with drug abuse, long term alcoholism that may impact the results of the trial;
10. Women during pregnancy or lactation, or fertile women unwilling to take contraceptive measures;
11. Non-appropriate patients for the trial according to the judgment of the investigators;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival（PFS） | up to 2 years
  Time from treatment until disease progression or death

SECONDARY OUTCOMES:
overall survival（OS） | up to 2 years
  Time from treatment until death from any cause
Treatment-related adverse events (AEs) | 2 years
  Physiological parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No